CLINICAL TRIAL: NCT05425771
Title: ARMA (Antireflux Mucosa Ablation) in Patients With Chronic Refractory Reflux Disease
Acronym: ARMA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Klinikum Garmisch-Patenkirchen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ARMA01
Record Dates: First submitted 2022-01-28; First posted 2022-06-21 (Actual); Last update posted 2022-07-14 (Actual); Status verified 2022-07

CONDITIONS: Gastro-esophageal Reflux; Reflux, Gastroesophageal
Keywords: Reflux disease; Endoscopic therapy
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Intervention Model Description: Pilot study of mucosal ablation for therapy refractory reflux disease
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mucosa Ablation Arm (Experimental): Treatment group
  Interventions: Procedure: Anti Reflux Mucosa Ablation

INTERVENTIONS:
Procedure: Anti Reflux Mucosa Ablation — Mucosa ablation with Argon plasma coagulation performed in inversion at the gastroesophageal junction in a crescent or horseshoe shape over a width of 1.5 - 2 cm in patients with refractory reflux symptoms

SUMMARY:
Pilot study of the possible clinical response to anti reflux mucosal ablation in patients with chronic refractory reflux disease

DETAILED DESCRIPTION:
Prospective, non-controlled, monocentric pilot study in patients with therapy-refractory reflux symptoms under proton pump inhibitor (PPI) therapy or intolerance of the necessary therapy or rapid recurrence of the symptoms with tapering therapy.

The symptoms must have existed for >6 months. Gastroesophageal reflux disease (GERD) must be diagnosed before inclusion in the study. This is the case if either erosive reflux esophagitis according to Los Angeles classification grades A-D is present or non-erosive reflux disease (NERD) has been confirmed by a 24-hour pH measurement/impedance measurement. The measurement must show either an increased number of reflux events or a prolonged time under reflux. In addition, there must be a high correlation between symptoms and reflux events when reporting symptom events. The GERD-HRQL score is queried for the clinical quantification of symptoms.

An esophageal motility disorder, especially achalasia or relevant hypomotility must be ruled out in an high resolution esophageal manometry. A relevant gastric emptying disorder is ruled out using a C13 octanoate breath test.

Patients with a Hill IV axial hernia, a paraesophageal hernia, or Barrett's esophagus are not included. Pregnancy must be ruled out in women of childbearing age.

The ARMA procedure is explained to the patient in detail with the expected benefits and risks in oral and written form. In addition, alternative treatments such as surgical fundoplication are discussed.

In the ARMA procedure, a gastroscopy is performed under sedation with propofol. Argon plasma coagulation (APC) is performed in inversion at the gastroesophageal junction in a crescent or horseshoe shape over a width of 1.5 - 2 cm, as described in the original publication. The intended destruction of the uppermost layer of the gastroesophageal junction is intended to induce an inflammatory reaction with subsequent shrinkage of the corresponding tissue section. This leads to a tightening of the gastroesophageal junction with subsequent improved tightness, so that reflux events occur less frequently.

Patients will be monitored in hospital for 48 hours. The existing drug therapy is continued for 4 weeks and then tapered off.

Endoscopic and clinical follow-up checks take place after 2 and 6 months using gastroscopy and GERD-HRQL score.

ELIGIBILITY:
Inclusion Criteria:

* typical reflux symptoms more than 2x per week during PPI therapy more than 6 month
* proof of gastro-esophageal reflux in pH metry oder pH/Impedance measurement

Exclusion Criteria:

* age < 18 y
* primary motility disorder of the esophagus
* hiatal hernia > 3 cm
* Hill classification > III
* pregnancy
* coagulation disorder
* mandatory intake of oral anticoagulation drugs

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2022-07-14 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-05-31 (Estimated)

PRIMARY OUTCOMES:
change of GERD-HRQL | Before and after 2 and 6 Month
  The Gastroesophageal Reflux Disease-Health Related Quality of Life (GERD-HRQL) is a standardized questionaire and a quantitative method of measuring symptom severity in gastroesophageal reflux disease (GERD). The results are from minimal 0 points up to 50 points. The higher the points, the greater the complaints.
Rate of major complications | day 1
  Recording of all major complication which require hospitalization

SECONDARY OUTCOMES:
Technical success nominal scale | Day 1
  In this case, the abortion of the procedure or the subjective assessment of the examiner apply immediately after the end of the procedure.
  The examiner evaluates the complete technical success as successful or unsuccessful
change of DeMeester Score | Before and after 2 and 6 Month
  The DeMeester score is a scoring system at pH/Impendence measurement that quantifies esophageal acid exposure time in long-term pH monitoring. A DeMeester score of ≤ 14.72 is considered physiological.
  The score includes the following values:
  Percentage of time with esophageal pH < 4 of total measurement time Percentage of time with pH < 4 during the waking phase (upright position) Percentage of time with pH < 4 during the sleep phase (lying position) Total number of reflux episodes during the measurement time Number of reflux episodes lasting > 5 min Duration of the longest reflux episode
change of reflux events | Before and after 2 and 6 Month
  Measurement of the number of events in the pH/Impendence measurement. A count <74 in 24 hours is considered normal.

CONTACTS AND LOCATIONS:
Locations (1):
- Klinikum Garmisch-Partenkirchen, Garmisch-Partenkirchen, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No